CLINICAL TRIAL: NCT00194688
Title: Breath Ammonia Method for H. Pylori Detection: Phase II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: David Kearney, MD, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 01-8470-V 04; 2R44DK055935-02 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Helicobacter Infections
Keywords: ammonia
MeSH Terms: conditions — Helicobacter Infections

INTERVENTIONS:
Drug: H. pylori treatment

SUMMARY:
The objective is to evaluate the utility of a breath ammonia sensing device. In this study we will assess the effect of H. pylori infection on breath ammonia levels by measuring whether there is a change in the pattern or quantity of breath ammonia seen in H. pylori positive patients compared to H. pylori negative patients.

DETAILED DESCRIPTION:
Healthy volunteers will undergo testing for H. pylori infection using a 14-C urea breath test, and the results will be compared to an experimental ammonia breath test. The breath sample will be collected by an investigational device that the patient will be exposed to consisting of a plastic mouth-piece which is attached to a T-tubing section having a side-arm port through which a fiberoptic ammonia sensor is inserted inside the tube. To meet the Phase II specific aim, the scope of the clinical trials is expanded addressing the following specific objectives:

* Test refinements of the sensing system (hardware, software, & breath test device)
* Determine whether a urea dose-response effect exists following urea ingestion,
* Define the optimal cutoff values for expired breath ammonia to allow optimal discrimination of H. pylori infected vs. uninfected persons.
* Determine the appropriate time interval for breath ammonia testing following urea ingestion.
* Determine whether there is a change in breath ammonia level after H. pylori treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers not meeting exclusion criteria

Exclusion Criteria:

* Known cirrhosis of the liver
* Renal insufficiency (BUN greater than 40 mg/dl, Creatinine greater than 2.0 mg/dl).
* Prior gastric resection
* Severe chronic obstructive pulmonary disease (Forced expiratory volume in 1 second less than 1.5 L)
* Patients unwilling or unable to discontinue proton pump inhibitors for 2 weeks prior to scheduled 14C or non-isotopic urea breath testing
* Patients who have received antibiotics or bismuth within the preceding month.
* Patients unwilling or unable to give informed consent
* Pregnant women (14C urea breath test is not approved for use in pregnant women)
* Age less than 21 years (14C urea breath test is not approved for use in children)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278
Dates: Start 2003-03; Study Completion 2005-06

PRIMARY OUTCOMES:
Sensitivity and specificity of breath ammonia measurement for H. pylori infection

SECONDARY OUTCOMES:
Determination of a dose response relationship for oral urea dose and breath ammonia level.
Determination of whether breath ammonia measurement allows determination of successful H. pylori treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David L Putnam, PhD, Study Director — Pacific Technologies, Inc.
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States